CLINICAL TRIAL: NCT05426434
Title: Intermittent Preventive Treatment in Pregnancy With Sulfadoxine-pyrimethamine Plus Dihydroartemisinin-piperaquine to Prevent Malaria Infection and Reduce Adverse Pregnancy Outcomes in Papua New Guinea - a Randomised Controlled Trial
Brief Title: Sulfadoxine-pyrimethamine Plus Dihydroartemisinin-piperaquine for Intermittent Preventive Treatment in Pregnancy
Acronym: SAPOT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Menzies School of Health Research (Other)
Collaborators: Papua New Guinea Institute of Medical Research (Other Government); University of Melbourne (Other); Curtin University (Other); Liverpool School of Tropical Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2021-4107
Record Dates: First submitted 2022-06-14; First posted 2022-06-22 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Malaria; Malaria in Pregnancy; Pregnancy Related
MeSH Terms: conditions — Malaria | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Intervention Model Description: Double blinded randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Placebos will be used to mimic the identical dosing strategy such that every 4 weeks women will receive two drugs on day 1 (SP and placebo, or SP and DP) followed by one drug on days 2 and 3 (placebo or DP). One placebo that mimics the appearance of DP will be used. A randomization list will be computer generated by a member of the project who will not be directly involved in the conduct of the study. The randomization list will include consecutive treatment numbers with corresponding random treatment assignments. Randomized codes will correspond to the 2 treatment arms using permuted variable sized blocks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SP + DP placebo every 4 weeks (Active Comparator): Control arm
  Interventions: Drug: Sulfadoxine pyrimethamine (SP)
- SP + DP given every 4 weeks (Experimental): Intervention arm
  Interventions: Drug: Dihydroartemisinin-Piperaquine (DP); Drug: Sulfadoxine pyrimethamine (SP)

INTERVENTIONS:
Drug: Dihydroartemisinin-Piperaquine (DP) — DP (D-Artepp) will be supplied by Fosun Pharma, China. DP will consist of three 40mg/320mg) tablets given once a day for three consecutive days
  Other Names: D-Artepp
  Arms: SP + DP given every 4 weeks
Drug: Sulfadoxine pyrimethamine (SP) — SP (G-COSPE) will be supplied by Fosun Pharma, China. SP will be given as a single dose consisting of three 500mg/25mg tablets.
  Other Names: G-COSPE

SUMMARY:
This trial tests the hypothesis that intermittent preventive treatment in pregnancy (IPTp) with sulfadoxine-pyrimethamine (SP) plus dihydroartemisinin-piperaquine (DP) significantly reduces the risk of malaria infection (primary outcome) and adverse birth outcomes (key secondary outcome) in an endemic area of Papua New Guinea (PNG), compared to IPTp with SP alone (the current standard of care).

To test this hypothesis a double-blinded, placebo-controlled, phase-III, superiority trial will individually randomize 1,172 HIV-uninfected pregnant women enrolled from 12-26 gestational weeks in equal proportions to one of two IPTp arms: 1) SP given every for weeks, or 2) SP+DP given every 4 weeks. DP placebos will be used to ensure adequate blinding is achieved in the study and follow-up will end 28 days after giving birth.

DETAILED DESCRIPTION:
Plasmodium falciparum and P. vivax infections cause malaria, maternal anemia and interfere with the development of the fetus, thereby increasing the risks of adverse pregnancy outcomes such as miscarriage, stillbirth, premature birth, fetal growth restriction, low birth weight, and infant death. Infected pregnant women are frequently asymptomatic, and current point-of-care tests miss placental and low-density infections. Monthly intermittent preventive treatment in pregnancy (IPTp) with sulfadoxine-pyrimethamine (SP) is designed to clear asymptomatic infections and provide post-treatment prophylaxis. The World Health Organization recommends IPTp with SP and long-lasting insecticidal bed nets for the prevention of malaria in pregnancy in endemic areas of sub-Saharan Africa. However, the emergence and spread of high-grade parasite resistance to SP threatens to compromise this strategy. Dihydroartemisinin-piperaquine (DP) is a safe fixed-dose artemisinin-based combination therapy used for the management of uncomplicated P. falciparum and P. vivax malaria in pregnancy and has emerged as a potential candidate to replace SP for IPTp. In comparative trials conducted in high-transmission settings in sub-Saharan Africa IPTp with DP was safe and significantly reduced the risk of P. falciparum infection compared to IPTp with SP. IPTp with DP also reduced the risk of P. vivax parasitemia in Papua Indonesia when compared to a single screen and treat approach. However, DP's superior antimalarial efficacy in African studies did not translate to large reductions in adverse pregnancy outcomes in these trials. This suggests that SP, whilst failing as an antimalarial, may prevent adverse pregnancy events via potent non-malarial effects that are not inherent to DP. For example, SP may provide protection from pathogens other than malaria parasites that are directly or indirectly involved in the causation of adverse pregnancy outcomes.

Papua New Guinea (PNG) is characterized by moderate intensity co-transmission of P. falciparum and P. vivax and a high burden of adverse pregnancy outcomes. PNG is the only country outside of Africa that has a policy of IPTp with SP. However, P. vivax resistance to SP is now common, high-grade P. falciparum resistance to SP may be emerging, and DP could provide enhanced antimalarial protection. However, given the high burden of adverse pregnancy outcomes from malaria- and non-malaria related causes, simply replacing SP with DP for IPTp in PNG may not lead to a reduction in adverse birth outcomes. Instead, combining DP with SP for IPTp has the potential to substantially improve health outcomes by reducing the risk of malaria infection whilst harnessing the non-malaria-related benefits of SP.

A double-blinded randomized controlled clinical trial will (1) compare the risk of malaria infection among pregnant women randomized to receive monthly IPTp with SP vs. SP+DP; (2) compare the risk of adverse pregnancy outcomes among pregnant women randomized to receive monthly IPTp with SP vs. SP+DP; and (3) compare safety and tolerability of monthly IPTp with SP vs SP+DP. The findings of this trial may have important policy implications, and the evidence generated will inform practice for PNG and sub-Saharan Africa.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 12-26 weeks' gestation
* 16 years of age or older
* Viable singleton intrauterine pregnancy
* Permanent resident of the study area
* Willing to adhere to scheduled and unscheduled study visit procedures
* Willing to birth in a study clinic or hospital
* Able to provide written informed consent

Exclusion Criteria:

* Multiple pregnancy (i.e. twins/triplets)
* Known heart ailment or other chronic medical condition requiring frequent hospital care
* Active medical problem requiring inpatient evaluation at the time of screening
* Severe malformations or non-viable pregnancy if observed by ultrasound
* Antimalarial therapy in the prior two weeks
* Unable to provide written informed consent
* Known allergy or contraindication to any of the study drugs
* Early or active labour
* Known HIV-positive status

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1172 (Estimated)
Dates: Start 2022-08-31 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Malaria infection in pregnancy | Starting two weeks after initial dose until and including delivery
  'Malaria infection in pregnancy' is a composite outcome, defined as one or more episode of P. falciparum and/or P. vivax infection, detected by microscopy and/or qPCR in peripheral blood or placental blood, or P. falciparum and/or P. vivax infection, detected as active infection on placental histology. The surveillance period will run from two weeks after the first dose of the first monthly treatment up until and including delivery (numerator) in women who attend at least one scheduled or unscheduled visit during the surveillance period (denominator).
  Proportion of women with 'malaria infection in pregnancy'

SECONDARY OUTCOMES:
Adverse pregnancy outcome | Time of delivery up to 28 days postpartum
  Composite adverse birth outcome is defined as the occurrence of any of the following:
  * Spontaneous miscarriage: Fetal loss <28 weeks of gestational age
  * Stillbirth: Infant born deceased at ≥28 weeks of gestational age
  * Low birth weight (LBW): Live birth with birth weight <2,500 grams
  * Preterm birth (PTB): Live birth <37 weeks gestational age
  * Small-for-gestational age (SGA): Live birth with birth weight-for-gestational-age <10th percentile of the INTERGROWTH-21st reference
  * Neonatal death: Live birth with neonatal death within the first 28 days of life
  Prevalence of adverse pregnancy outcome
Clinical malaria during pregnancy | Starting two weeks after initial dose until and including delivery
  Incidence of new episodes of fever or history of fever plus positive RDT confirmed by microscopy and/or qPCR during pregnancy
Parasitemia during pregnancy | Starting two weeks after initial dose until and including delivery
  Proportion of samples with parasites detected in maternal peripheral blood samples by microscopy or qPCR
Composite placental malaria detected by microscopy, qPCR or by histology | At time of delivery
  Prevalence of placental parasites by microscopy, qPCR, or placental histology
Placental malaria detected by microscopy | At time of delivery
  Prevalence of parasites in placental blood by microscopy
Placental malaria detected by qPCR | At time of delivery
  Prevalence of parasites in placental blood by qPCR
Active placental malaria detected by histology | At time of delivery
  Prevalence of active infection (presence of parasites) on histology
Past placental malaria detected by histology | At time of delivery
  Prevalence of past infection (pigment only) on histology
Placental malaria detected by histology | At time of delivery
  Prevalence of placental infection (active or past) on histology
Composite fetal loss and neonatal death | Time of delivery up to 28 days postpartum
  Prevalence of fetal loss (spontaneous miscarriage or stillbirth) and neonatal death
Composite of SGA-LBW-PTB | At time of delivery
  Prevalence of small for gestational age, low birth weight, and preterm birth
SGA | At time of delivery
  Prevalence of small for gestational age using the new Intergrowth-21st population reference's 10th centile
LBW | At time of delivery
  Prevalence of low birth weight
PTB | At time of delivery
  Prevalence of preterm birth
Birth weight | At time of delivery
  Mean birthweight
Neonatal length | At time of delivery
  Neonatal length
Maternal nutritional status | 8 months from randomisation
  Changes in maternal body mass index (BMI)
Maternal nutritional status | 6 months from randomisation
  Changes in maternal mid-upper arm circumference (MUAC)
Maternal anemia during pregnancy and at delivery | 6 months from randomisation
  Proportion of routine haemoglobin measurements <100 g/L
Maternal hemoglobin levels during pregnancy and at delivery | 6 months from randomisation
  Mean hemoglobin (g/L) at the third trimester antenatal visit and at delivery
Congenital anemia | At delivery
  Prevalence of anaemia (Hb <130 g/L) from newborn cord blood
Maternal gametocyte carriage during pregnancy and at delivery | 6 months from randomisation
  Proportion of P. falciparum positive samples with gametocytes at the third trimester antenatal visit and at delivery, by light microscopy and RT-qPCR
Molecular markers of DP resistance | 6 months from randomisation
  Proportion of parasite positive samples with molecular markers of DP resistance
Molecular markers of SP drug resistance | 6 months from randomisation
  Proportion of parasite positive samples with molecular markers of SP resistance
Maternal mortality | 8 months from randomisation
  he death of a woman while pregnant or within 42 days of the end of pregnancy, irrespective of the duration and site of the pregnancy, but not from accidental or incidental causes
Congenital malformations | 8 months from randomisation
  Any visible external congenital abnormality on surface examination
Other SAEs and AEs | 8 months from randomisation
  Incidence of AEs and SAEs
(History) of vomiting study drug | 6 months from randomisation
  Prevalence of vomiting investigational product (IP) twice at the same IP administration visit
Dizziness | 6 months from randomisation
  Prevalence of dizziness after a course of IP
Gastrointestinal complaints | 6 months from randomisation
  Prevalence of gastrointestinal complaints after a course of IP

CONTACTS AND LOCATIONS:
Overall Officials: Holger Unger, PhD MBChB, Principal Investigator — Menzies School of Health Research, Darwin, Australia
Locations (1):
- Papua New Guinea Institute of Medical Research, Madang, Madang Province, Papua New Guinea

IPD SHARING:
Plan to Share IPD: No